CLINICAL TRIAL: NCT01991639
Title: Nutrition Intervention and Physical Training in Malnourished, Frail, Community-dwelling, Elderly Subjects Carried Out by Trained Lay "Buddies"
Brief Title: Healthy Life for Frail Malnourished Seniors Performed Together With Trained Lay Buddies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Priv. Doz. Thomas E. Dorner, Priv. Doz, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12-039
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Frail Elderly; Malnutrition
Keywords: frailty; community-dwelling; malnutrition; physical activity; nutritional intervention
MeSH Terms: conditions — Malnutrition; Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive training (No Intervention): Participants are visited twice a week by buddies, but they do not specifically monitor the nutritional status or perform physical training in the first 10-12 weeks. Instead of that buddies are provided with a portfolio of possible activities, especially cognitive training, which they could perform together with the frail, malnourished subjects.
- nutritional & physical activity (Experimental): Buddies visit malnourished, frail, elderly subjects twice a week for approximately one hour and they perform nutritional and physical activity interventions.
  Interventions: Other: Nutritional and physical activity intervention

INTERVENTIONS:
Other: Nutritional and physical activity intervention — Buddies visit malnourished, frail, elderly subjects twice a week for approximately one hour and they perform nutritional and physical activity interventions.
  Arms: nutritional & physical activity

SUMMARY:
Background: In elderly subjects frailty and malnutrition are very common and can lead to serious health hazards, increase mortality, morbidity, dependency, institutionalization and a reduced quality of life. In Austria, the prevalence of frailty and malnutrition are increasing steadily and are becoming a challenge for our social system. Physical training and adequate nutrition can invert it.

Methods/Design: In this randomized, controlled trial 80 malnourished, frail, community-dwelling patients (≥ 65 years) are recruited. Additionally, 80 lay volunteers (≥ 50 years) named buddies are recruited and subsequently trained regarding health enhancing physical activity and nutrition in three standardized training sessions. These buddies visit the malnourished, frail subjects at home twice a week for about one hour during an initial period of 10-12 weeks. While participants allocated to the intervention group (n=40) conduct intervention to improve their fluid intake, their protein and energy intake, perform strength training and try to increase their baseline activities, the control group (n=40) only gets home visits without any special intervention. After 10-12 weeks, both, the intervention and the control group, receive the nutrition intervention and the physical training. Health, nutrition and frailty status, physical fitness and body composition and chronic inflammation of buddies and frails are recorded before the intervention, after 10-12 weeks, and after 6 and 12 months.

Discussion: To the investigators knowledge this trial is the first of its kind to provide nutrition and physical activity intervention to malnourished, frail, community-dwelling subjects by trained lay buddies, in which the health status of buddies is also expected to improve. This study assesses the effectiveness of such an intervention. If successful, the intervention offers new perspectives for the management of frailty and malnutrition.

ELIGIBILITY:
Inclusion Criteria frail, malnourished subjects:

* 65 years or older
* Living in Vienna
* Hospital discharged planned for the next 14 days
* Malnutrition or at risk of malnutrition according to the MNA-SF
* Frail or pre-frail according to the SHARE-FI
* Community-dwelling
* No medical contraindication for the performance of physical strength training
* Able to walk (with or without a walking aid)
* Capability to consent

Exclusion Criteria frail, malnourished subjects:

* 65 years or younger
* Admission to nursing home is planned
* Nursing level 6 or 7
* Cancer according to the medical charts
* Insulin treated diabetes mellitus according to the medical charts
* COPD stage III or IV
* Dialysis patient
* Cannot understand the German language
* Impaired cognitive function according to the MMSE (≤ 17 points)

Inclusion Criteria buddies:

* 50 years or older
* Signed informed consent
* Readiness to participate in the study as well in the intervention as in the control group
* Commitment to keep to the protocol for at least 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in handgrip at 10-12 weeks and at 6 and 12 months | Before the intervention, after 10-12 weeks and after 6 and 12 months

SECONDARY OUTCOMES:
Change from baseline in nutritional status at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Risk for malnutrition is assessed by the long form of the mini nutritional assessment (MNA).
Change from baseline is frailty status at 10-12 weeks and at 6 and 12 months | Before the intervention, after 10 -12 weeks and after 6 and 12 months
  For the assessment of frailty the SHARE-FI as used in the Survey of Health, Ageing and Retirement in Europe will be applied.
Change from baseline in quality of life at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Quality of life is assessed by the WHOQOL-BREF and by 3 dimensions of the WHOQOL-OLD ("sensory functions", "autonomy", "activities in the past, present and future".
Changes from baseline in social support at 10-12 weeks and at 6 months | before the intervention, after 10-12 weeks and after 6 months
  The social support is assessed by the Fragebogen zur sozialen Unterstützung (FSozU K-14).
Changes from baseline in sings of malnutrition and frailty at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks, and after 6 months
  Laboratory parameters (albumin, total cholesterol, transferrin, triglyceride, 25-hydroxy-vitamin D, folic acid, CRP, IL-6, TNF-alpha and leucocytes)
Changes from baseline in cognitiv function at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Cognitiv function is assessed by the Mini Mental State Examination (MMSE).
Changes from baseline in muscle strength after 10-12 weeks and 6 months | Before the intervention, after 10 -12 weeks and after 6 months
  Muscle strength is assessed by the MASS (Measurement of age and sex related reference values of muscle strength) and the Concept dyno 2. The MASS is a new diagnosis system which was developed by the Technical University of Vienna. It evaluates health related concentric dynamic muscle strength. The measurement is velocity-independent and hence, is appropriate for the target group. Three exercises (bench press, bench pull, and leg press) will be conducted in standardized procedure. For all tested muscle groups the following parameters are recorded: maximum resistance with low velocity and 2-3 fix adjusted sub-maximum loads. Moreover, the Concept 2 dyno is used for assessing the muscle strength. The same exercises as before will be conducted in standardized procedure and the results are analyzed according to the reference values
Changes from baseline in the amount of physical activity at 10-12 weeks and 6 months | Before the intervention, after 10-12 weeks and after 6 months
  The amount of physical activity is assessed by the Physical Activity Scale for the Elderly (PASE) and a modified version of the FEG (Fragebogen zur Erfassung des Gesundheitsverhaltens).
  Moreover each patient receives a pedometer to measure the daily steps.
Changes from baseline in balance and mobility components at 10-12 weeks and at 6 months | Before the intervenion, after 10-12 weeks and after 6 months
  The Short Physical Performance Battery (SPPB) is a method for assessing physical performance of older patients.
Changes from baseline in qualitative and quantitative contents of refrigerator at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Predefined protocol of the refrigerator of the frail individuals will assess the refrigerator contents which will be classified as adequate, inadequate (rotten food or just beyond the date stamped on the label), or empty (less than three different food products)
Changes from baseline in quality of the whole diet at 10-12 week and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Changes in the quality of the whole diet is assesseb by Mediterranean Diet Adherence Screener (MEDIAS), a food frequency questionnaire assessing the protein intake and questions concerning supplements
Measures of drop-out after 10-12 weeks | Afer 10-12 weeks
Measures of adherence after 10 -12 weeks | after 10 -12 weeks
Appraisal of the participant after 10-12 weeks | after 10-12 weeks
Documentation of any undesirable event during the intervention after 6 months | after 6 months
Changes from baseline in frequency of hospitalization at 10-12 weeks and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
Changes from baseline in frequency of falls at 10-12 weeks and 6 months | Before the intervention, after 10-12 weeks and after 6 months
Changes from baseline in fear of fallings at 10-12 week and at 6 months | Before the intervention, after 10-12 weeks and after 6 months
  Falls Efficacy Scale International (FES-I) was developed for the documentation of fall-related self-efficacy in older persons by an EU-funded expert network (Prevention of Falls Network Europe ProFaNE)
Measures of drop-out after 6 months | Afer 6 months
Measures of adherence after 6 months | after 6 months
Expectations of the participant before the intervention | Before the intervention
Appraisal of the participant after 6 months | after 6 months
Documentation of any undesirable event during the intervention after 10-12 weeks | after 10 -12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Dorner, Priv.Doz., Principal Investigator — Institut für Sozialmedizin
Locations (1):
- Institute of Social Medicine, Centre for Public Health, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lackinger C, Grabovac I, Haider S, Kapan A, Winzer E, Stein KV, Dorner TE. Adherence Is More Than Just Being Present: Example of a Lay-Led Home-Based Programme with Physical Exercise, Nutritional Improvement and Social Support, in Prefrail and Frail Community-Dwelling Older Adults. Int J Environ Res Public Health. 2021 Apr 15;18(8):4192. doi: 10.3390/ijerph18084192. PMID 33920981
- [Derived] Grabovac I, Haider S, Winzer E, Kapan A, Schindler KE, Lackinger C, Dorner TE. Changes in health parameters in older lay volunteers who delivered a lifestyle-based program to frail older people at home. Wien Klin Wochenschr. 2018 Nov;130(21-22):637-644. doi: 10.1007/s00508-018-1372-6. Epub 2018 Aug 9. PMID 30094663
- [Derived] Kapan A, Winzer E, Haider S, Titze S, Schindler K, Lackinger C, Dorner TE. Impact of a lay-led home-based intervention programme on quality of life in community-dwelling pre-frail and frail older adults: a randomized controlled trial. BMC Geriatr. 2017 Jul 19;17(1):154. doi: 10.1186/s12877-017-0548-7. PMID 28724351
- [Derived] Dorner TE, Lackinger C, Haider S, Luger E, Kapan A, Luger M, Schindler KE. Nutritional intervention and physical training in malnourished frail community-dwelling elderly persons carried out by trained lay "buddies": study protocol of a randomized controlled trial. BMC Public Health. 2013 Dec 27;13:1232. doi: 10.1186/1471-2458-13-1232. PMID 24369785